CLINICAL TRIAL: NCT02019485
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess Bioequivalence of a New Tapentadol Extended-Release (TRF) 100-mg Tablet With Respect to a Tapentadol Extended-Release (PR2) 100-mg Tablet Under Fasted Conditions in Healthy Subjects
Brief Title: A Study to Assess Bioequivalence of a New Tapentadol Extended-Release Tablet With Respect to a Tapentadol Extended Release Tablet Under Fasted Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100457; R331333-PAI-1060 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); HP5503/83 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Healthy; Tapentadol; Tapentadol extended-release tamper-resistant formulation; Tapentadol extended-release prolonged-release formulation; Bioequivalence; Fasted Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive single dose of new tapentadol Extended Release (ER) Tamper-Resistant Formulation (TRF) tablet and later, participants will receive single dose of current tapentadol prolonged-release formulation 2 (PR2) tablet without food. Administration of the study medications will be separated by a washout period (no treatment) of 7 to 14 days.
  Interventions: Drug: Tapentadol Extended Release (ER) Tamper-Resistant Formulation (TRF); Drug: Tapentadol Prolonged-Release Formulation 2 (PR2)
- Treatment Sequence BA (Experimental): Participants will receive single dose of current tapentadol PR2 tablet and later, participants will receive single dose of new tapentadol ER TRF tablet without food. Administration of the study medication will be separated by a washout period of 7 to 14 days.
  Interventions: Drug: Tapentadol Extended Release (ER) Tamper-Resistant Formulation (TRF); Drug: Tapentadol Prolonged-Release Formulation 2 (PR2)

INTERVENTIONS:
Drug: Tapentadol Extended Release (ER) Tamper-Resistant Formulation (TRF) — Participants will receive a single dose of tapentadol ER TRF 100 mg tablet orally (by mouth) in treatment sequences AB and BA appropriately.
Drug: Tapentadol Prolonged-Release Formulation 2 (PR2) — Participants will receive a single dose of tapentadol PR2 100 mg tablet orally in treatment sequences AB and BA appropriately.

SUMMARY:
The purpose of this study is to evaluate bioequivalence (biological equivalence of two formulations of a study medication) of a new tapentadol Extended release (ER) 100 mg tamper-resistant formulation (TRF) tablet, to the current tapentadol ER 100 mg, prolonged-release formulation 2 (PR2) tablet used in healthy participants under fasted (without food) conditions.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), 2-way crossover (method used to switch participants from one treatment arm to another in a clinical study), single-dose, and single-center study. The study consists of 3 phases: the screening phase, treatment phase, and end-of-study or withdrawal assessment phase. In the treatment phase, participants will receive a single dose of new tapentadol ER 100-mg TRF tablet (Treatment A) and current tapentadol ER 100-mg PR2 (Treatment B) under fasted conditions in 2 treatment sequences (AB and BA). Administration of the study medication will be separated by a washout period (no treatment) of 7 to14 days. Approximately 64 participants will be enrolled in this study. Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination. The duration of participation in the study for an individual participant will be approximately 5.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to protocol-defined use of effective contraception
* Body mass index (BMI) between 20 and 28 kilograms per square meter, inclusive, and body weight not less than 50 kg (BMI is calculated as weight [kilogram] divided by square of height [meter])
* Habitually smokes no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before the first study medication administration

Exclusion Criteria:

* History of seizure disorder or epilepsy or mild or severe traumatic brain injury
* Men with hemoglobin concentrations below 12.5 g/dL or women with hemoglobin concentrations below 11.5 g/dL
* Positive test for drugs of abuse, such as cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, or barbiturates at screening or Day -1 of each treatment period
* Positive test for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies
* History of a gastrointestinal disease affecting absorption, gastric surgery or history of or current significant medical illness

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration of tapentadol | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication)
Time to reach the observed maximum serum concentration of tapentadol | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Area under the serum concentration-time curve of tapentadol from time 0 to the time of the last quantifiable concentration | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Area under the serum concentration-time curve of tapentadol from time 0 to infinite time | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Percentage of area under the serum concentration-time curve of tapentadol from time 0 to infinite time | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Elimination half-life associated with the terminal slope of the semilogarithmic tapentadol concentration-time curve | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
First-order rate constant associated with the terminal portion of tapentadol concentration curve | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Time to last quantifiable serum concentration of tapentadol | Predose; 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, and 48 hours postdose (at each single-dose of study medication
Number of participants with adverse events | Up to end-of-study (Day 3 of last single-dose of study medication)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Lincoln, Nebraska, United States